CLINICAL TRIAL: NCT04931745
Title: Virtual Reality for Procedural Distress in Children Undergoing Port-a-Cath Access: A Randomized Controlled Trial
Brief Title: Virtual Reality for Port-a-Cath Access
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 119117
Record Dates: First submitted 2021-05-14; First posted 2021-06-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Oncology Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality (Experimental): The Oculus 2 headset will be used during port access. The device features a stereoscopic display mounted on a lightweight wireless head mounted display weighing 503 g with built-in 3D audio and an adjustable head strap and adjustable lens distance. The software used will be the Might Pebbles VR Game developed by ManageXR. It is a child-friendly VR game that does not require the use of hand controllers. It also provides an option to increase the cognitive load, making it appropriate for children of all ages. The experimental group will be given up to 10 minutes to familiarize themselves with the device, assisted by the research assistant and will begin using it 5-10 minutes prior to port access. Most participants will receive topical anesthestic in the form of 4% amethocaine (Ametop), eutectic mixture of lidocaine and amethocaine (EMLA), or 4% lidocaine (Maxilene) as per standard practice at our institution. However, some participants may refuse this co-intervention.
  Interventions: Device: Virtual reality
- Tablet (Active Comparator): The child will watch a video on a tablet or iPad that is appropriate for their age during port access. They will begin using it 5-10 minutes prior to port access. The content of the video will be at the discretion of the child life specialist, nurse, or caregiver. Most participants will receive topical anesthestic in the form of 4% amethocaine (Ametop), eutectic mixture of lidocaine and amethocaine (EMLA), or 4% lidocaine (Maxilene) as per standard practice at our institution. However, some participants may refuse this co-intervention.
  Interventions: Device: Tables distraction
- No or non-technologic distraction (Active Comparator): This is no distraction or non-technologic distraction measures such as bubbles, etc., facilitated by the child life specialist, nurse, or caregiver during port access. The measure will be documented for the purposes of analysis. They will begin using it 5-10 minutes prior to port access. Most participants will receive topical anesthestic in the form of 4% amethocaine (Ametop), eutectic mixture of lidocaine and amethocaine (EMLA), or 4% lidocaine (Maxilene) as per standard practice at our institution. However, some participants may refuse this co-intervention.
  Interventions: Other: No or non-technologic distraction

INTERVENTIONS:
Device: Virtual reality — VR headset will be used 5-10 minutes prior to and during port access
  Other Names: Oculus 2
  Arms: Virtual Reality
Device: Tables distraction — Tablet distraction will be used 5-10 minutes prior to and during port access
  Other Names: iPad
  Arms: Tablet
Other: No or non-technologic distraction — This approach will be used 5-10 minutes prior to and during port access
  Arms: No or non-technologic distraction

SUMMARY:
Children with cancer almost universally receive port-a-catheters (ports) to deliver medication, fluids, blood products, and conduct blood tests. Port access requires a needle inserted through the skin to the subcutaneous tissue. Despite the application of topical anesthetic, port access can be painful and anxiety producing. Virtual reality (VR) interfaces provide a strategy to reduce anxiety and have been employed in other painful procedures in children. This trial will explore the effectiveness of VR in children undergoing port access.

DETAILED DESCRIPTION:
Pain management in pediatric oncology patients is a core component of the care provided. Procedures and treatment administration are the greatest sources of pain for these children, often greater than the pain from the disease itself. Poor initial management for procedures can lead to anxiety and fear, along with a heightened pain response for future procedures. Sensitization, which is an increased reaction to pain, may not only occur at a physiological level, but can also psychologically affect these children, resulting in the development of a fear-avoidance response. This can impede the conduct of diagnostic testing and delivery of therapy. It can also result in an overall fear and avoidance of healthcare settings.

Port-a-caths are a medical device that is implanted below the skin, which acts as a type of venous access. They are used in pediatric oncology patients for various reasons including administration of chemotherapeutics, blood products and supportive care medication, venous sampling and diagnostic testing. At our centre, 90% of patients have a port, while the 10% remaining either have a Hickman catheter or PICC line. Acute lymphoblastic leukemia (ALL), has a treatment duration of two and half years which is facilitated by the insertion of a port-a-cath. To access a port, the area is cleaned in a sterile fashion and a needle is inserted through the skin, into the port. Ports must be flushed with heparin for line maintenance every 4-6 weeks. Currently, topical analgesics such as EMLA (lidocaine/prilocaine), and distraction methods such as interactive toys and watching videos, and anticipatory guidance are employed to help decrease the amount of pain and anxiety children encounter while their port is accessed5,6. Although topical analgesia and child life interventions may decrease the amount of procedural pain and distress, they do not fully eliminate it. Virtual Reality (VR) has been commercially available for almost 25 years, but the initially high cost prohibited widespread clinical adoption. It is being explored as a potential form of analgesia, and has been found to be effective at decreasing pain in numerous settings including in pediatric burn patients undergoing dressing changes, outpatient venipuncture, and port-cath access. The mechanism by which VR works to reduce pain is still unclear, but it has been suggested that it is through distraction. Studies using functional MRI have also shown that VR reduces pain-associated brain activity. For some children, the use of topical agents prolongs the period of distress in anticipation of port access, something, which the use of VR may diminish/eliminate.

Given that VR technology is still quite new, there have been limited studies in the use of VR in port-a-cath access. Sample sizes of previous studies investigating the use of VR in port-a-cath access have been small, ranging between 20 to 59 patients. Additional limitations include the use of non-objective, self-report and proxy measures of distress, use of a non-active comparator (no intervention), and the lack of young children (< 7 years). However, port-a-cath access is common in young children and is often more distressing. Further, for some children the use of topical agents for access creates/prolongs period of distress to do anticipation of port-a-cath access. Behavioral measures of distress are more accurate than self-report and proxy measures. Standards of care to reduce procedural distress usually involves some type of distraction too. To optimize the external generalizability of our findings, the investigators have designed a trial to overcome these limitations, including a larger sample size, an objective measure of behavioral distress, inclusion of younger children, and an active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Children age 5 to 17 years of age who are undergoing port-a-cath access
* Pre-intervention Children's Fear Scale score of at least 1 with respect to the impending port-a-cath access

Exclusion Criteria:

* Subjective report of motion sickness within past 12 months (excluding anticipatory nausea a child may experience en route to their medical appointment)
* Subjective history of claustrophobia Requires timely antimicrobial therapy
* Visual, auditory, or cognitive impairment or language barrier precluding comprehension of study-related tasks or safe interaction with VR
* Medical record documentation of current MRSA infection
* Subjective history of concurrent respiratory infection (defined as cough, sore throat, fever, coryza, or sneezing within the past 24 hours) or gastrointestinal infection (defined as any vomiting or diarrhea within past 24 hours)
* Previous enrollment in study
* Seizure disorder
* History of vertigo or neurological disorder that creates moderate to severe dizziness.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Behavioral distress | During intervention
  The Observational Scale of Behavioral Distress - Revised (OSBD-R) will be used. The OSBD-R is an 8-factor, weighted observational scale with total scores ranging between 0 to 23.5 (0 = no distress, 23.5 = maximal distress) , validated in children 1 to 20 years of age for measuring distress associated with medical procedures. This will be measured at the first attempt at port access.

SECONDARY OUTCOMES:
Pain Intensity | During intervention
  Pain intensity will be measured using the Faces Pain Scale - Revised (FPS-R) immediately following port-a-cath access and reflective of the pain experienced during port access. The Faces Pain Scale is a self-reported measure that uses 6 faces to assess the intensity of children's pain26. It has been validated in children as young as 4 years of age and has a strong positive correlation with the visual analogue scale (r = 0.93 in children 5-12 years of age; r = 0.92 in children 4-12 years of age) and the colour analogue scale (r = 0.84 in children 4-12 years old). It conforms closely to a linear rating scale.
Fear | During intervention
  Measured using the Children Fear Scale (CFS) immediately following port-a-cath access and reflective of fear felt during port access. The Children's Fear Scale is a visual scale validated to measure fear in children as young as 5 years old undergoing a painful medical procedure. It was originally validated in children undergoing venipuncture and showed interrater reliability of 0.51, test-retest reliability of 0.76, convergent validity with another self-report measure of fear of 0.73, and moderate discriminant validity of 0.30 with child coping behaviour and 0.41 with child distress behaviour.
Immersiveness | During intervention
  Measured using the Child Presence Measure (CPM) immediately after port access and reflective of their experience with the VR intervention. This outcome will only be obtained from the participants in the VR group. It has been shown that immersive virtual environments decreases the subjective experience of pain. The Child Presence Measure is a 12-question survey that measures immersiveness of the VR experience.
Frequency of adverse events | During intervention
  These will include but are not limited to:
  1. Nausea using the Pediatric Nausea Assessment Tool (PeNAT). The PeNAT is an assessment tool for nausea validated for children undergoing chemotherapy, which uses a standardized script for administration and employs a pictorial scale.
  2. Vomiting
  3. Dizziness Adverse events will be recorded as those that occur from the initial application of the intervention to 15 minutes post intervention

OTHER OUTCOMES:
Parental distress | During intervention
  Measured using the Parental Distress Questionnaire (PDQ) immediately following port access and reflective of distress felt related to port-a-cath access. The Parental Distress Questionnaire is a self-reported survey where parents are given 4 emotional adjectives reflecting emotional distress, which are rated on an 11-point numeric scale ranging from 0 = "not at all" to 11 = "extremely" to assess the parent's current distress.
Need for physical restraint during port access | During intervention
  Yes or no
Number of port-a-cath access attempts | During intervention
Length of stay | During intervention
  Measured from initial nursing assessment to discharge
Duration of port-a-cath access procedure | During intervention
  Measured from removal of topical anesthetic (if any) to attempted flush of port.
Procedure nurse satisfaction with intervention | During intervention
  Measured from the procedure nurse using the VR Distraction Satisfaction Questionnaire.
  This Questionnaire was developed by Stinson et al. to measure ease of needle insertion, acceptability of VR intervention use, helpfulness of VR intervention, and impact of VR intervention on clinical work flow (nurses' report). It uses a 5-point Likert scale from "unacceptable" to "very acceptable" for nurses.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No